CLINICAL TRIAL: NCT06314880
Title: A Phase I, Single Center, Randomized, Double-blind, Placebo-controlled Study to Evaluation the Safety, Tolerability, and Immunogenicity of Recombinant Meningococcal Group B Vaccine (E.Coli) in a Population Aged 3 Months-50 Years Old
Brief Title: Safety, Tolerability, and Immunogenicity of Recombinant Meningococcal Group B Vaccine (E.Coli)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022112701
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: Recombinant Meningococcal Group B Vaccine (E. Coli)
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 18-50 years old (Experimental): 60 people per age group. The first 15 subjects in the 18-50 age group will serve as sentinels, with 10 in the experimental group and 5 in the control group.
  Interventions: Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (low-dose); Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (hign-dose); Biological: Placebo control
- 6-17 years old (Experimental): 60 people per age group. Divided into high-dose group, low-dose group, and placebo group.
  Interventions: Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (low-dose); Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (hign-dose); Biological: Placebo control
- 2-5 years old (Experimental): 60 people per age group. Divided into high-dose group, low-dose group, and placebo group.
  Interventions: Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (low-dose); Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (hign-dose); Biological: Placebo control
- 6-23 months old (Experimental): 60 people per age group. Divided into high-dose group, low-dose group, and placebo group.
  Interventions: Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (low-dose); Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (hign-dose); Biological: Placebo control
- 3-5 months old (Experimental): 60 people per age group. Divided into high-dose group, low-dose group, and placebo group.
  Interventions: Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (low-dose); Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (hign-dose); Biological: Placebo control

INTERVENTIONS:
Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (low-dose) — Each dose contains 60μg of MenB-fHBP-A and MenB-fHBP-B respectively. Administer one dose of 0.5mL each time. 20 people/group.
Biological: Recombinant Meningococcal Group B Vaccine (E. Coli) (hign-dose) — Each dose contains 100μg of MenB-fHBP-A and MenB-fHBP-B respectively. Administer one dose of 0.5mL each time. 20 people/group.
Biological: Placebo control — Placebo control. 20 people/group.

SUMMARY:
The research objective is to evaluate the safety and tolerability of the recombinant Group B meningococcal vaccine (E. coli) and explore its preliminary immunogenicity.

DETAILED DESCRIPTION:
This is a Phase I, single center, randomized, double-blind, placebo-controlled clinical trial conducted in Guangxi Province, China. The purpose of this study is to evaluate the safety and tolerability of the recombinant Group B meningococcal vaccine (E. coli) and explore its preliminary immunogenicity. Expected to include 300 subjects, divide them into 5 age groups of 18-50 years old, 6-17 years old, 2-5 years old, 6-23 months old, and 3-5 months old, and 2 dose groups, a total of 10 groups, with 30 people in each group. The experimental group and placebo control group are 20 people and 10 people, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 3 months to 50 years old, legal guardian and/or individual can provide legal identification;
* The subjects and/or their legal guardians have the ability to understand the research procedures, agree to participate in the study (and/or their legal guardians agree to the child's participation in the study), and sign an informed consent form;
* The subjects and/or their legal guardians are able to participate in all planned follow-up visits;
* On the day of enrollment, the axillary temperature was less than 37.3 ℃;
* Standards for certain groups of people:
* Subjects ≥ 2 years old: laboratory test indicators (as specified in the protocol) within the normal range, or those with abnormalities but no clinical significance (evaluated by clinical doctors);
* Female participants of childbearing age: Agree to take effective contraceptive measures within 6 months from enrollment to full vaccination.

Exclusion Criteria:

* Have received any Group B meningococcal vaccine in the past;
* A history of invasive diseases caused by meningococcus or gonococci;
* Pregnant or lactating women;
* Have any history of severe allergies to vaccines or drugs in the past, such as allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura;
* Suffering from serious heart disease, liver disease, kidney disease, congenital malformations, developmental disorders, and genetic defects (including but not limited to Down syndrome, moderate to severe thalassemia, etc.) that may interfere with the progress or completion of the study;
* Diagnosed as having congenital or acquired immunodeficiency, or suspected of having serious chronic or systemic diseases that may interfere with the conduct or completion of the study, such as active tuberculosis, hepatitis B, hepatitis C, human immunodeficiency virus (HIV), syphilis infection, etc;
* Individuals with encephalopathy, uncontrolled epilepsy, seizures, and other progressive neurological disorders, or a history or family history of mental illness;
* Suffering from contraindications for intramuscular injection such as thrombocytopenia, any coagulation disorders, or receiving anticoagulant therapy;
* Received immunosuppressive therapy within 3 months prior to vaccination, such as continuous use of systemic glucocorticoid therapy for more than 2 weeks, such as prednisone or similar drugs>5mg/day (note: local and inhaled/nebulized steroids can be used);
* Asplenia or splenectomy, functional asplenia caused by any circumstances;
* Subjects with hypertension (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg, suitable for adults);
* Suffering from acute illness or in the acute phase of chronic illness, or using antipyretic, analgesic, and antiallergic drugs (such as acetaminophen, ibuprofen, aspirin, etc.) three days before the first dose of vaccination;
* Within 7 days (≤ 7 days) prior to enrollment, received inactivated vaccines, and within 14 days (≤ 14 days) received live attenuated vaccines;
* Has received blood or blood related products or immunoglobulin (hepatitis B immunoglobulin is acceptable) within 3 months prior to enrollment;
* Premature infants (gestational age<37 weeks), low birth weight infants (birth weight<2500g), and infants with a history of abnormal labor (only applicable to the 3-5 month and 6-23 month age groups);
* Plan to move before the end of the study or leave the local area for a long time during the scheduled study visit;
* Participating in or planning to participate in clinical trials of other drugs in the near future;
* The researchers believe that there are any conditions in the subjects that may interfere with the evaluation of the research objectives.

Ages: 3 Months to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-07-22 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of all AEs within 0-30 days after each dose of vaccination | within 0-30 days after vaccination
  All AEs occurrence within 0-30 days after each dose of vaccination (occurrences, number of cases, incidence rate, and relationship with vaccination)
The incidence rate of solicited AEs within 30 minutes after each dose of vaccination | within 30 minutes after vaccination
  All solicited AEs occurrence within 30 minutes after each dose of vaccination (occurrences, number of cases, incidence rate, and relationship with vaccination)
The incidence rate of solicited AEs within 0-14 days after each dose of vaccination | within 0-14 days vaccination
  All solicited AEs occurrence within 0-14 days after each dose of vaccination (occurrences, number of cases, incidence rate, and relationship with vaccination)
The incidence rate of unsolicited AEs within 0-30 days after each dose of vaccination | within 0-30 days vaccination
  All unsolicited AEs occurrence within 0-30 days after each dose of vaccination (occurrences, number of cases, incidence rate, and relationship with vaccination)
The incidence rate of grade 3 and higher AEs within 0-30 days after each dose of vaccination | within 0-30 days vaccination
  All grade 3 and higher AEs occurrence within 0-30 days after each dose of vaccination (occurrences, number of cases, incidence rate, and relationship with vaccination)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Nanning, Guangxi, China